CLINICAL TRIAL: NCT04624165
Title: Patient Perspective of Telemedicine in Gynecology Oncology
Status: Completed | Type: Observational
Sponsor: TriHealth Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 20-092
Record Dates: First submitted 2020-10-26; First posted 2020-11-10 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-08

CONDITIONS: Oncology
Keywords: Telemedicine
MeSH Terms: conditions — Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — o We plan to hand out copies of a survey to examine patient's perspective on telemedicine.

SUMMARY:
Research question: do patients in a gynecologic oncology practice value the use of telemedicine as an adjunct to in-person visits and in what circumstances might patients not find these visits to be sufficient?

DETAILED DESCRIPTION:
In the United States, 14.8 million women live greater than 50 miles away from the closest gynecology oncologist underscoring the need for increased implementation of telemedicine. In consideration of the COVID-19 outbreak, recommendations were made to organize goals of therapy by prioritizing curative intent and utilizing telemedicine to manage current therapies. Research regarding telemedicine, its benefits, and patient perspectives in other specialties has been reported, however there appears to be a dearth of information in the field of gynecologic oncology. Our study aims to seek patients' perspective of telemedicine and whether implementation for extended office visits, teleconsultations and more are feasible and valuable to them.

ELIGIBILITY:
o Eligible patients would be at least 18 years of age, and currently being treated by one of the providers within the gynecologic oncology group.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: o Eligible patients would be at least 18 years of age, and currently being treated by one of the providers within the gynecologic oncology group.
Sampling Method: Non-Probability Sample
Enrollment: 116 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Patient's perspective on telemedicine on a Likert Scale | Through survey completion, an average of 15 minutes
  Patient's perspective on telemedicine on a Likert Scale

CONTACTS AND LOCATIONS:
Overall Officials: Robert Neff, MD, Principal Investigator — TriHealth Inc.
Locations (1):
- TriHealth - Good Samaritan and Bethesda North Hospitals, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No